CLINICAL TRIAL: NCT01053364
Title: Feasibility Study of NL-Prow Interspinous Spacer Device and Procedure
Brief Title: Feasibility Study of NL-Prow Interspinous Spacer to Treat Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Non-Linear Technologies (Industry)
Responsible Party: Lilach Eyal / Clinical Manager, Non-Linear Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL-PROW-01
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

ARMS (1):
- Implant (Experimental)
  Interventions: Device: NL-Prow interspinous spacer implant

INTERVENTIONS:
Device: NL-Prow interspinous spacer implant — Interspinous spacer implant

SUMMARY:
The purpose of the study is to evaluate the clinical safety and feasibility of the NL-Prow™ Interspinous Spacer implant and insertion procedure in the treatment of lumbar spinal stenosis

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥50 years of age.
* Symptoms of leg/buttock/groin pain, with or without back pain, that are exacerbated by lumbar extension and relieved in flexion.
* Diagnosis of neurogenic intermittent claudication (NIC) (defined as a feeling of paresthesia and/or discomfort and/or pain and/or weakness in the leg(s) during walking or standing) secondary to lumbar spinal canal stenosis at 1-2 lumbar levels (between L1 and L5), confirmed by dynamic X-Ray (showing sagital instability or rocking), and CT and/or MRI (showing central spinal canal narrowing and/or foraminal narrowing).
* Has completed at least 6 months of conservative therapy, which may include but is not limited to, epidural steroid injections, oral steroids, NSAIDS, analgesics, physical therapy, spinal manipulation, bracing.
* Appropriate candidate for lumbar surgical treatment using posterior approach.
* Subject can walk independently 15 meters or more.
* Subject is able to understand the risks and benefits of participating in the study.
* Subject understands and has signed the study informed consent form.
* Subject is physically and mentally willing and able to comply with the requirements of the study procedure and scheduled follow-up visits and testing.

Exclusion Criteria:

* Severe symptomatic lumbar spinal stenosis at ≥2 level, requiring surgical intervention.
* Prior lumbar spine surgery at any level.
* Unremitting pain in any spinal position or axial back pain only without leg/buttock/groin pain.
* Evidence that subject's symptoms are due to vascular claudication OR has significant peripheral vascular disease.
* Significant instability of the lumbar spine at any level OR defined as translation of more than 3mm or 10 degrees of angular motion between flexion and extension on upright lateral radiographs.
* Subject has an ankylosed segment at the affected level.
* Significant scoliosis, defined as Cobb angle >25°.
* Cauda equina syndrome.
* Fixed motor deficit or known peripheral neuropathy demonstrated clinically.
* Subject has degenerative neurologic disease.
* Subject has any mass lesions.
* Any evidence of spinal or systemic infection.
* Subject has a history of spinous process fracture or pars interarticularis fractures or pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips
* Subject has history or radiographic evidence of 1 or more osteoporotic fractures in the spine.
* Subject has severe osteoporosis of the spine, defined as bone mineral density (BMD) in the spine more than 2.5 SD below the mean of adult normals.
* Subject is paraparetic.
* Subject has a bleeding disorder.
* Active systemic disease such as HIV, hepatitis, etc.
* Subject is immunologically suppressed, or has received or is receiving 7.5 milligrams prednisone (or equivalent) daily for more than six months immediately prior to enrollment.
* Extreme morbid obesity, defined as BMI >35 kg/m2.
* Diagnosis of lumbar spinal stenosis which requires a direct neural decompression or surgical intervention other than those required to implant the experimental device.
* Subject is not able to undergo MRI or tolerate closed MRI scan.
* Known or suspected history of alcohol and/or drug abuse.
* Life expectancy less than one year.
* Active rheumatoid arthritis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Accurate placement of the interspinous spacer confirmed by fluoroscopy | Procedure completion

SECONDARY OUTCOMES:
Improvement in leg and or back pain and in walking capability compared to baseline | One year
Any device and or procedure related adverse events or complications | One year

CONTACTS AND LOCATIONS:
Overall Officials: Zdenek Novak, MD, PhD, Principal Investigator — St. Anne's University Hospital Brno, Czech Republic
Locations (1):
- Neurosurgery department, St. Anne's University Hospital, Brno, Czechia